CLINICAL TRIAL: NCT00508651
Title: An Expanded Phase1/2a Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Immunogenicity, and Viral Shedding of MEDI-560, A Live, Attenuated Recombinant Parainfluenza Virus Type 3 (PIV3) Vaccine, Administered Intranasally to Healthy Infants 1 to <12 Mos. of Age
Brief Title: A Phase 1/2A Study to Evaluate the Safety, Immunogenicity, and Shedding of MEDI-560 in Infants 1 to < 12 Months of Age
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was closed prior to enrollment of Cohort 2 due to a non-safety related sponsor decision.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Judith Falloon , MD, MedImmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP150; NCT01150799 (obsolete NCT alias)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Results first posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: parainfluenza virus, children, vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 MEDI-560 (Experimental): MEDI-560 vaccine was a frozen preparation of live, attenuated rHPIV3cp45 virus filled into Becton Dickinson^TM Luer slip tip syringes. Each 0.2 mL dose contained 10^5 TCID50 of MEDI-560 in a sucrose phosphate glutamate buffer.
  Interventions: Biological: MEDI-560
- Cohort 1 Placebo (Placebo Comparator): Placebo was a frozen preparation filled into Becton Dickinson^TM Luer slip-tip syringes. Each 0.2 mL dose contained sucrose phosphate buffer.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MEDI-560 — MEDI-560 vaccine was a frozen preparation of live, attenuated rHPIV3cp45 virus filled into Becton Dickinson^TM luer slip tip syringes. Each 0.2 mL dose contained 10^5 TCID50 of MEDI-560 in a sucrose phosphate glutamate buffer.
  Arms: Cohort 1 MEDI-560
Biological: Placebo — Placebo was a frozen preparation filled into Becton Dickinson^TM luer slip-tip syringes. Each 0.2 mL dose contained sucrose phosphate buffer.
  Arms: Cohort 1 Placebo

SUMMARY:
The primary objective of this study is to describe the safety and tolerability of 3 doses of MEDI-560 at 10^5 TCID50 when administered to children 6 to < 12 months of age who are HPIV3 (human parainfluenza virus type 3) seronegative at baseline and to infants 1 to < 3 months of age regardless of baseline serostatus.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multidose Phase 1/2a multicenter study designed to evaluate the safety, tolerability, viral shedding, immunogenicity, and genotypic and phenotypic stability of MEDI-560 in infants 1 to < 12 months of age. Three doses of MEDI-560 at a dosage level of 10^5 TCID50 were administered 0, 2, and 4 months after enrollment to a 30-participant cohort of 6 to < 12 month-old HPIV3 seronegative children randomized 2:1 to MEDI-560 vs placebo. A second 160-participant cohort of 1 to < 3 month-old infants not screened for baseline serostatus was planned but was not opened to enrollment for reasons other than safety. Participants were followed for safety through 180 days post last dose. Nasal wash specimens were collected at screening and Days 7, 12, and 28 following each dose and during unscheduled illness visits to assess vaccine virus shedding and genotypic and phenotypic stability of any shed vaccine virus. Blood was collected at screening to determine eligibility and prior to Dose 1 for baseline serostatus. Blood for assessment of antibodies to HPIV3 was collected approximately 7 to 12 days after Dose 1 and Dose 3 and 1 month after each dose for antibodies to PIV3.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female whose age on the day of randomization falls within one of the two age cohorts:

   Cohort 1: 6 to < 12 months (≥ 6 months of age and not yet reached their 1st year birthday); Cohort 2: 1 to < 3 months (> 28 days of age and not yet reached their 3rd month birthday)
2. Cohort 1 only: Participant is seronegative to HPIV3 at screening as determined by ELISA; or the legal representative is willing to provide access to data documenting that the participant was screened for another MedImmune trial after written informed consent was obtained, and that the participant is seronegative to HPIV3 within 21 days prior to randomization into MI-CP150 as determined by ELISA at MedImmune
3. Participant was the product of a normal full term pregnancy, defined as 36-42 weeks gestation
4. Participant is in general good health
5. Participant's legal representative is available by telephone
6. Written informed consent and Health Insurance Portability and Accountability Act authorization (if applicable) obtained from the participant's legal representative
7. Participant's legal representative is able to understand and comply with the requirements of the protocol as judged by the investigator
8. Participant is available to complete the follow-up period of 180 days after the final dose of investigational product as required by the protocol
9. Participant's legal representative is willing and able to bring the subject to the study site for evaluation of respiratory illness in accordance with the protocol

Exclusion Criteria:

1. Any fever (≥ 100.4°F [≥ 38.0°C], regardless of route) or lower respiratory illness within 7 days prior to randomization
2. Moderate or severe nasal congestion that in the investigator's opinion could prevent intranasal delivery of investigational product
3. Cohort 1 only: weight < the fifth percentile for age on the day of randomization
4. Cohort 2 only: history of low birth-weight (ie, < 2,500 grams at birth) or weight < fifth percentile for age on the day of randomization
5. Any drug therapy (chronic or other) within 7 days prior to randomization or expected receipt through the protocol-specified blood collection 28 days after each investigational product dosing, except that infrequent use of over-the-counter medications such as pain relievers are permitted according to the judgment of the investigator
6. Any current or expected receipt of immunosuppressive agents including steroids (≥ 2 mg/kg per day of prednisone or its equivalent, or ≥ 20 mg/day if the participant weighs >10 kg, given daily or on alternate days for ≥ 14 days); children in this category should not receive investigational product until immunosuppressive agents including corticosteroid therapy have been discontinued for ≥ 30 days; the use of topical steroids is permitted according to the judgment of the investigator
7. History of receipt of blood transfusion or expected receipt through 30 days after final investigational product dosing
8. History of receipt of immunoglobulin products or expected receipt through 30 days after final investigational product dosing
9. Receipt of any investigational drug within 60 days prior to randomization or expected receipt through 30 days after final investigational product dosing
10. Receipt of any live virus vaccine (excluding rotavirus vaccine) within 28 days prior to randomization or expected receipt within a 28-day window around any dose
11. Receipt of any inactivated (eg, non-live) vaccine or rotavirus vaccine within 14 days prior to randomization or expected receipt within a 14-day window around any dose
12. Known or suspected immunodeficiency, including human immunodeficiency virus
13. Living in the same home or enrolled in the same classroom at day care with infants < 24 months of age within 28 days after each dose (only one child per household may be enrolled into the study)
14. Contact with pregnant caregiver within 28 days after each dose
15. Household contact with an immunocompromised person within 28 days after each dose; the participant should also avoid close contact with immunocompromised individuals for at least 28 days after each investigational product dose
16. Household contact within 28 days after each dose with a healthcare worker who has direct patient care responsibilities or household contact within 28 days after each dose with someone who is a day care provider or preschool teacher for children < 24 months of age
17. History of allergic reaction to any component of the investigational product
18. Previous medical history or evidence of an intercurrent or chronic illness that, in the opinion of the investigator, may compromise the safety of the participant
19. Known or suspected active or chronic hepatitis infection
20. History of medical diagnosis of asthma, reactive airway disease, wheezing requiring medication, bronchoconstriction or treatment with a β2 agonist (eg, albuterol), cystic fibrosis, chronic lung disease of prematurity (eg, bronchopulmonary dysplasia), chronic pulmonary disease, medically confirmed apnea, hospitalization for respiratory illness or mechanical ventilation
21. A family member or a household contact who is an employee of the research center or otherwise involved with the conduct of the study
22. Any condition that, in the opinion of the investigator, might interfere with investigational product evaluation

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Falloon, MD, Study Director — MedImmune LLC
Locations (23):
- United States (23):
  - Children's Investigational Research Program, Bentonville, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Madera Family Medical Group, Madera, California
  - Allergy Medical Group of the North Area, Roseville, California
  - Miami Children's Hospital, Miami, Florida
  - Homestead Clinical Research, Naranja, Florida
  - University of South Florida College of Medicine Department of Pediatrics, Tampa, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Michael W. Simon, M.D., Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - Children's Lung Specialists Ltd., Las Vegas, Nevada
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke Health Center- Pickett Road, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Belleview Pediactric Assoc., Pittsburgh, Pennsylvania
  - Holston Medical Group, Kingsport, Tennessee
  - Dixie Pediatrics, St. George, Utah
  - University Physicians Internal Medicine, Huntington, West Virginia

REFERENCES:
- [Result] Bernstein DI, Falloon J, Yi T. A randomized, double-blind, placebo-controlled, phase 1/2a study of the safety and immunogenicity of a live, attenuated human parainfluenza virus type 3 vaccine in healthy infants. Vaccine. 2011 Sep 16;29(40):7042-8. doi: 10.1016/j.vaccine.2011.07.031. Epub 2011 Jul 22. PMID 21782874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 6 to < 12 months of age were screened prior to randomization at 8 sites in the USA. The first and last days of informed consent were 07Nov2007 and 30Jun2008, respectively. No participants were screened for Cohort 2 (1 to < 3 months of age) because the study was closed prior to enrollment into Cohort 2 for reasons other than safety.
Pre-assignment Details: Thirty participants were randomized into Cohort 1 between 12Nov2007 and 07Jul2008. Participants were randomized in a 2:1 ratio to receive MEDI-560 or placebo, and randomization into Cohort 1 was not stratified.
Groups:
- Cohort 1 MEDI-560: MEDI-560 vaccine was a frozen preparation of live, attenuated rHPIV3cp45 virus filled into Becton Dickinson™ Luer slip tip syringes. Each 0.2 mL dose contained 10^5 TCID50 of MEDI 560 in a sucrose phosphate glutamate buffer.
- Cohort 1 Placebo: Placebo was a frozen preparation filled into Becton Dickinson™ Luer slip-tip syringes. Each 0.2 mL dose contained sucrose phosphate buffer.
Period: Overall Study
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Started | 20 | 10
Completed | 16 | 8
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age Continuous [Mean (Standard Deviation); unit: Months] | 8.94 (1.85) | 8.44 (1.20) | 8.77 (1.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (SEs) After Dose 1
Time Frame: Days 0-28 after Dose 1 (Dose 1 was on Day 0)
Population: Safety population for solicited symptoms included randomized participants who received investigational product for the specified dose and had any solicited symptom data obtained after that dose
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participants
  runny/stuffy nose | 14 | 6
  cough | 13 | 5
  drowsiness | 8 | 2
  irritability/fussiness | 6 | 2
  fever greater than or equal to 100.4° F | 3 | 1
  fever greater than or equal to 101.5° F | 1 | 0
  fever greater than or equal to 103.2° F | 1 | 0
  fever greater than or equal to 104.9° F | 0 | 0
  loss of appetite/decreased urine output | 3 | 2
  oropharygeal inflammation (laryngitis) | 1 | 0
  epistaxis | 0 | 0

2. Primary Outcome: Number of Participants With SEs After Dose 2
Time Frame: Days 0-28 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 6
participants
  runny/stuffy nose | 12 | 4
  cough | 6 | 2
  drowsiness | 3 | 0
  irritability/fussiness | 8 | 2
  fever greater than or equal to 100.4° F | 5 | 1
  fever greater than or equal to 101.5° F | 2 | 1
  fever greater than or equal to 103.2° F | 1 | 0
  fever greater than or equal to 104.9° F | 0 | 0
  loss of appetite/decreased urine output | 4 | 0
  oropharygeal inflammation (laryngitis) | 2 | 0
  epistaxis | 0 | 0

3. Primary Outcome: Number of Participants With SEs After Dose 3
Time Frame: Days 0-28 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 7
participants
  runny/stuffy nose | 7 | 3
  cough | 5 | 1
  drowsiness | 2 | 0
  irritability/fussiness | 6 | 3
  fever greater than or equal to 100.4° F | 3 | 0
  fever greater than or equal to 101.5° F | 2 | 0
  fever greater than or equal to 103.2° F | 0 | 0
  fever greater than or equal to 104.9° F | 0 | 0
  loss of appetite/decreased urine output | 4 | 1
  oropharygeal inflammation (laryngitis) | 0 | 0
  epistaxis | 0 | 0

4. Primary Outcome: Number of Participants With Adverse Events (AEs) After Dose 1
Description: Unsolicited AEs reported by 1 or more participants in either treatment group through 28 days post Dose 1.
Time Frame: Days 0-28 after Dose 1 (Dose 1 was on Day 0)
Population: Safety population for adverse events included randomized participants who received investigational product for the specified dose and had any safety follow-up after that dose (ie, did not discontinue on Day 0 after that dose).
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participants
  Tachycardia | 2 | 0
  Conjunctivitis | 1 | 0
  Diarrhoea | 3 | 1
  Vomiting | 2 | 1
  Gastroenteritis | 1 | 0
  Otitis media | 3 | 0
  Upper respiratory infection | 5 | 2
  Body temperature increased | 1 | 0
  Pharyngeal erythema | 1 | 0
  Rhinorrhea | 2 | 1
  Dermatitis atopic | 1 | 0
  Rash | 0 | 1

5. Primary Outcome: Number of Participants With AEs After Dose 2
Description: Unsolicited AEs reported by 1 or more participants in either treatment group through 28 days post Dose 2.
Time Frame: Days 0-28 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 6
participants
  Conjunctivitis | 2 | 0
  Diarrhoea | 2 | 0
  Vomiting | 1 | 0
  Gastroenteritis | 1 | 1
  Otitis media | 1 | 0
  Upper respiratory infection | 8 | 2
  Body temperature increased | 2 | 0
  Pharyngeal erythema | 1 | 0
  Rhinorrhea | 0 | 1
  Dermatitis atopic | 0 | 1
  Rash | 1 | 2

6. Primary Outcome: Number of Participants With AEs After Dose 3
Description: Unsolicited AEs reported by 1 or more participants in either treatment group through 28 days post Dose 3.
Time Frame: Days 0-28 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 7
participants
  Conjunctivitis | 1 | 0
  Diarrhoea | 2 | 2
  Vomiting | 1 | 0
  Otitis media | 1 | 0
  Upper respiratory infection | 2 | 1
  Body temperature increased | 1 | 0
  Dermatitis atopic | 0 | 1
  Rash | 0 | 1

7. Primary Outcome: Number of Participants With Medically Attended Lower Respiratory Illnesses (MA-LRIs) After Dose 1
Time Frame: Days 0-28 after Dose 1 (Dose 1 was on Day 0)
Population: Safety population for MA-LRIs included randomized participants who received investigational product for the specified dose and had any safety follow-up after that dose (ie, did not discontinue on Day 0 after that dose)
Measure: Number; unit: participant
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participant
  Bronchiolitis | 1 | 0
  Wheezing | 1 | 0
  Pneumonia | 0 | 0

8. Primary Outcome: Number of Participants With MA-LRIs After Dose 2
Time Frame: Days 0-28 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 7
Measure: Number; unit: participant
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 6
participant
  Bronchiolitis | 0 | 0
  Wheezing | 0 | 0
  Pneumonia | 1 | 0

9. Primary Outcome: Number of Participants With MA-LRIs After Dose 3
Time Frame: Days 0-28 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 7
Measure: Number; unit: participant
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 7
participant
  Bronchiolitis | 0 | 0
  Wheezing | 0 | 0
  Pneumonia | 0 | 0

10. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) After Dose 1
Time Frame: Days 0-28 after Dose 1 (Dose 1 was on Day 0)
Population: Safety population for SAEs included randomized participants who received investigational product for the specified dose and had any safety follow-up after that dose (ie, did not discontinue on Day 0 after that dose)
Measure: Number; unit: participant
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participant | 0 | 0

11. Primary Outcome: Number of Participants With SAEs After Dose 2
Description: One participant had event of pneumonia after Dose 2.
Time Frame: Days 0-28 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 6
participants | 1 | 0

12. Primary Outcome: Number of Participants With SAEs After Dose 3
Time Frame: Days 0-28 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 7
participants | 0 | 0

13. Primary Outcome: Number of Participants With Significant New Medical Conditions (SNMCs)
Description: A SNMC is a newly diagnosed medical condition that is of a chronic, ongoing nature and is assessed by the investigator as medically significant.
Time Frame: Day 0 through 180 days after final dose
Population: Safety population was randomized participants who received investigational product and had any safety follow-up, including a temperature measurement, SE, AE, concomitant medication use, or follow-up for ≥ 1 day after dosing (ie, did not discontinue on Day 0 after receiving Dose 1).
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participants | 0 | 0

14. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at Any Time During Study Participation
Description: Number of participants with nasal wash specimens that were culture positive for HPIV3 in which vaccine-like virus was identified.
Time Frame: Days 7, 12, and 28 after each dose and during visits for pre-specified illness symptoms occurring Day 0 through 180 days post final dose.
Population: The shedding population included all randomized participants who received investigational product and for whom at least one shedding sample result was available.
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participants | 17 | 0

15. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 7 Days After Dose 1
Description: as for outcome 14
Time Frame: Days 7-10 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participants | 16 | 0

16. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 12 Days After Dose 1
Description: as for outcome 14
Time Frame: Days 12-18 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 8
participants | 13 | 0

17. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 28 Days After Dose 1
Description: as for outcome 14
Time Frame: Days 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 7
participants | 0 | 0

18. Secondary Outcome: Number of Participants With Shedding of Vaccine-like Virus on Any Day During Days 0-28 After Dose 1
Time Frame: Days 0-34 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 20 | 8
participants | 17 | 0

19. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 7 Days After Dose 2
Description: as for outcome 14
Time Frame: Days 7-10 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 5
participants | 1 | 0

20. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 12 Days After Dose 2
Description: as for outcome 14
Time Frame: Days 12-18 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 18 | 6
participants | 0 | 0

21. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 28 Days After Dose 2
Description: as for outcome 14
Time Frame: Days 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 6
participants | 0 | 0

22. Secondary Outcome: Number of Participants With Shedding of Vaccine-like Virus on Any Day During Days 0-28 After Dose 2
Description: as for outcome 14
Time Frame: Days 0-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 19 | 6
participants | 1 | 0

23. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 7 Days After Dose 3
Description: as for outcome 14
Time Frame: Days 7-10 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 6
participants | 0 | 0

24. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 12 Days After Dose 3
Description: as for outcome 14
Time Frame: Days 12-18 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 15 | 7
participants | 0 | 0

25. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 28 Days After Dose 3
Description: as for outcome 14
Time Frame: Days 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 15 | 7
participants | 0 | 0

26. Secondary Outcome: Number of Participants With Shedding of Vaccine-like Virus on Any Day During Days 0-28 After Dose 3.
Description: as for outcome 14
Time Frame: Days 0-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 16 | 7
participants | 0 | 0

27. Secondary Outcome: Number of Participants With Hemagglutination Inhibition (HAI) Seroconversion/Seroresponse to HPIV3 28 Days After Dose 1
Description: Hemagglutination inhibition seroconversion/seroresponse is equal to or greater than a 4-fold rise in HAI antibody titer from baseline. Hemagglutination inhibition antibody results obtained on or after detection of wild-type HPIV3 in culture were not considered valid.
Time Frame: Days 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: The immunogenicity population included all randomized participants who received investigational product and who did not have a major protocol violation that would affect interpretation of immune response assay results and who had valid HAI results.
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 18 | 7
participants | 11 | 0

28. Secondary Outcome: Number of Participants With HAI Seroconversion/Seroresponse to HPIV3 28 Days After Dose 2
Description: as for outcome 27
Time Frame: Days 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 15 | 6
participants | 11 | 1

29. Secondary Outcome: Number of Participants With HAI Seroconversion/Seroresponse to HPIV3 28 Days After Dose 3
Description: as for outcome 27
Time Frame: Days 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 13 | 6
participants | 10 | 2

30. Secondary Outcome: Number of Nasal Wash Samples Containing Vaccine-like Virus in the Absence of Admixture With Wild-type HPIV3 in Which the Vaccine-like Virus Was Genotypically Stable
Description: A nasal wash specimen was collected at screening and on Days 7 (7-10), 12 (12-18), and 28 (28-34) post each dose and during visits for pre-specified illness symptoms occurring Day 0 through 180 days post final dose to assess vaccine virus replication. Genotypic stability of recovered vaccine-type virus at the 15 mutations of phenotypic importance was assessed.
Time Frame: Day 0 after Dose 1 to 180 days after the final dose
Population: All nasal wash samples in which MEDI-560 was identified in the absence of wild-type HPIV3 and for which valid genotype data are available
Measure: Number; unit: samples containing vaccine-like virus
Units Other Than Participants: nasal wash samples
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 17 | 0
Number analyzed (nasal wash samples) | 29 | 0
samples containing vaccine-like virus | 28 |

31. Secondary Outcome: Number of Nasal Wash Samples Containing Vaccine-like Virus in the Absence of Admixture With Wild-type HPIV3 in Which the Vaccine-like Virus Was Phenotypically Stable
Description: A nasal wash specimen was collected at screening and on Days 7 (7-10), 12 (12-18), and 28 (28-34) post each dose and during visits for pre-specified illness symptoms occurring Day 0 through 180 days post final dose to assess vaccine virus replication. Determination of the temperature sensitivity of recovered vaccine-type virus.
Time Frame: Day 0 after Dose 1 to 180 days after the final dose
Population: All nasal wash samples in which MEDI-560 was identified in the absence of wild-type HPIV3 and for which valid phenotype data are available
Measure: Number; unit: samples containing vaccine-like virus
Units Other Than Participants: Samples
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 17 | 0
Number analyzed (Samples) | 28 | 0
samples containing vaccine-like virus | 28 |

32. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Antibodies to HPIV3 at Baseline
Description: Pre-dose GMT of HAI antibody to HPIV3
Time Frame: Baseline (Day 0 prior to Dose 1)
Population: Immunogenicity population was randomized participants who received investigational product, did not have a protocol violation that would affect interpretation of immunogenicity results, and had valid HAI results. HAI results obtained on/after detection of wild-type HPIV3 were not considered valid. A value of 2 was assigned for HAI titers < 4.
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 18 | 6
GMT | 3.05 [2.2 to 4.8] | NA [NA to NA] — Results were less than the assay's limit of quantification, therefore were all imputed to be 2.0.

33. Secondary Outcome: Geometric Mean Titers of Serum Antibodies to HPIV3 Day 28 Post Dose 1
Description: Post-Dose 1 GMT of HAI antibody to HPIV3
Time Frame: Day 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 18 | 7
GMT | 17.28 [9.3 to 33.3] | NA [NA to NA] — Results were less than the assay's limit of quantification, therefore were all imputed to be 2.0.

34. Secondary Outcome: Geometric Mean Titers of Serum Antibodies to HPIV3 Day 28 Post Dose 2
Description: Post-Dose 2 GMT of HAI antibody to HPIV3
Time Frame: Day 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 15 | 6
GMT | 25.40 [11.1 to 55.7] | 3.17 [2.0 to 8.0]

35. Secondary Outcome: Geometric Mean Titers of Serum Antibodies to HPIV3 Day 28 Post Dose 3
Description: Post-Dose 3 GMT of HAI antibody to HPIV3
Time Frame: Day 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Number analyzed (Participants) | 13 | 6
GMT | 42.91 [13.3 to 142.4] | 6.35 [2.0 to 26.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 28-day period following each dose of investigational product. Serious adverse events were collected from Day 0 through 180 days after the final dose of investigational product.
Description: Other adverse events include events that occurred in at least 1 subject within 28 days after any dose.
Arm/Group | Cohort 1 MEDI-560 | Cohort 1 Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/8
Other Adverse Events (participants affected / at risk) | 19/20 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 MEDI-560 (N=20) | Cohort 1 Placebo (N=8)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 MEDI-560 (N=20) | Cohort 1 Placebo (N=8)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (4)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 4 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (15) | 4 (6)
Body temperature increased (Investigations) | 3 (4) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Cohort 2 was not enrolled due to a sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it is understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.